CLINICAL TRIAL: NCT05509322
Title: Care Expansion Across Remote Environments - Substudy of the SELF-GYN [Sonograms Enable Looking Forward - Get Your iNformation] Extension - I Trial
Brief Title: Care Expansion Across Remote Environments - Sub-Study of the SELF-GYN1 Trial
Acronym: CARE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is no longer going to be occurring- no subjects were enrolled at any point.
Sponsor: Turtle Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 016a
Record Dates: First submitted 2022-08-10; First posted 2022-08-22 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Fertility Risk

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, multi-arm real-world study
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded in the sense that they will be offered the consult at a particular price, and may be informed of the expected list price of the consult (i.e. what the price would be without the subsidy offered to the patient), but patients will not be aware that others are being offered different levels of subsidy.
  Independent raters will be blinded as to the level of subsidy the patient has received; reasonable effort will be made to maintain investigator blinding; however, nothing will prevent the patient from proactively mentioning to the investigator the price they are paying or considering paying for the consult.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Invitation to fertility consult with subsidy (Experimental): This group will be invited to purchase a fertility consult, and will be offered a subsidy if they choose to purchase the consult.
  Interventions: Other: Subsidy for fertility consult; Other: Invitation to purchase fertility consult
- Invitation to fertility consult without subsidy (Active Comparator): This group will be invited to purchase a fertility consult at full price.
  Interventions: Other: Invitation to purchase fertility consult
- Control (no invitation) (No Intervention): This group will not receive invitations to purchase a fertility consult.

INTERVENTIONS:
Other: Subsidy for fertility consult — Some participants will receive a subsidy when they purchase the fertility consult.
  Arms: Invitation to fertility consult with subsidy
Other: Invitation to purchase fertility consult — Some participants will receive an invitation from their health center to purchase an at-home fertility consult.
  Arms: Invitation to fertility consult with subsidy; Invitation to fertility consult without subsidy

SUMMARY:
This real-world, interventional sub-study will evaluate the impact of potential payer subsidies for Turtle Health at-home consults on subsequent interactions with the healthcare system within select sub-populations of interest.

DETAILED DESCRIPTION:
The present study is a sub-study of the SELF-GYN1 study. The SELF-GYN1 study is a multicenter study designed to evaluate the efficacy and safety of the use of the Turtle Health Ultrasound Scanner for the acquisition of transvaginal ultrasound images by a study participant, with no previous training, in her home when guided by real-time remote supervision from a qualified and specially trained ultrasound technologist.

In addition to the main questions of the SELF-GYN1 study, additional questions related to patient decision-making and pricing dynamics for patients who purchase patient's decisions to purchase a fertility consult alongside enrolling in the SELF-GYN1 trial, will be studied at Mayo Clinic, through providing subsidies for the purchasing of the fertility consult.

ELIGIBILITY:
Inclusion Criteria:

* All inclusion criteria from the SELF-GYN1 trial apply
* Participant in Mayo Clinic health system
* Lives in MN
* Belongs to a sub-population targeted for enrollment that has not yet met its enrollment target
* Consent to participate in electronic health record monitoring and outreach

Exclusion Criteria:

* All exclusion criteria from the SELF-GYN1 trial apply
* Planning to move away from MN in the next year

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Image quality | 6 weeks
  Percent of women whose stills are clinical quality, in each of 3 populations of interest.

SECONDARY OUTCOMES:
False positives | 6 weeks
  Rate of false positives of 'significant findings'
Recalled Net Promoter Score | 6 weeks
  Difference between recalled in-clinic Net Promoter Score and at-home Net Promoter Score. The Net Promoter Score has a range of 0-10 with higher scores indicating more favorable responses.
Number of patients opening box at correct time | 6 weeks
  Confirming patient opens box at correct time (not early)
Number of correct patients identified | 6 weeks
  Correct patient is identified by tech and tests (not wrong patient)
Number of patients who used probe cover | 6 weeks
  Patient correctly applies probe cover without either a) failing to apply it or b) ripping it, including in low light or other sub-optimal conditions
Number of patients placing probe in correct cavity | 6 weeks
  Patient places probe in correct cavity (vaginal vs. anal)
Rate of return packages sent | 6 weeks
  Patient ships product back in a timely fashion
Rate of probes that crack | 6 weeks
  Probe does not crack on out-return trip
Rate of working probes | 6 weeks
  Probe remains in working condition
Rate of probes being reprocessed | 6 weeks
  Probe is reprocessed properly per internal SOPs
Adverse events | 6 weeks
  Number and type of adverse events that occur
Number of participants per subsidy | 6 months
  Level of participation (purchase and completion of consult) per subsidy level within each cohort of interest
Number of couples who participate | 6 months
  Level of participation in couple consults where offered - i.e., purchase of both male and female consult, per subsidy level within each cohort of interest
Clinically significant findings | 6 weeks
  Percentage of patients in which clinically significant findings are identified
Number of IVF cycles | 6 months
  Number of IVF cycles conducted
Percentage of IVF cycles | 6 months
  Percentage of IVF cycles considered clinically necessary based on treating physician survey
Number of gynecological surgeries | 6 months
  Number of gynecological surgeries conducted
Percentage of minimally invasive gynecological surgeries | 6 months
  Percentage of those surgeries that are considered minimally invasive based on treating physician survey
Percentage of gynecological surgeries | 12 months
  Percentage of those surgeries that are considered clinically necessary within next 12 months based on treating physician survey
Number of additional TVUS | 6 months
  Number of additional transvaginal ultrasounds conducted to monitor findings identified during at-home consult
Number of other follow-up care | 6 months
  Number of other follow-up care sought based on findings identified during at-home consult
Percentage of follow up care per arm | 6 months
  Percentage of patients in each arm seeking follow up care of any kind; fertility care in particular after consult

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Chung EH, Petishnok LC, Conyers JM, Schimer DA, Vitek WS, Harris AL, Brown MA, Jolin JA, Karmon A, Styer AK. Virtual Compared With In-Clinic Transvaginal Ultrasonography for Ovarian Reserve Assessment. Obstet Gynecol. 2022 Apr 1;139(4):561-570. doi: 10.1097/AOG.0000000000004698. Epub 2022 Mar 10. PMID 35271530
- [Background] Birch Petersen K, Maltesen T, Forman JL, Sylvest R, Pinborg A, Larsen EC, Macklon KT, Nielsen HS, Hvidman HW, Nyboe Andersen A. The Fertility Assessment and Counseling Clinic - does the concept work? A prospective 2-year follow-up study of 519 women. Acta Obstet Gynecol Scand. 2017 Mar;96(3):313-325. doi: 10.1111/aogs.13081. Epub 2017 Feb 3. PMID 27990627
- [Background] Farquhar C, Ekeroma A, Furness S, Arroll B. A systematic review of transvaginal ultrasonography, sonohysterography and hysteroscopy for the investigation of abnormal uterine bleeding in premenopausal women. Acta Obstet Gynecol Scand. 2003 Jun;82(6):493-504. doi: 10.1034/j.1600-0412.2003.00191.x. PMID 12780419